CLINICAL TRIAL: NCT02768454
Title: Appropriate Use of Controlled Broad-spectrum Antimicrobials by Establish Stewardship and Execute by Antibiotic Pharmacist
Brief Title: Antimicrobials Stewardship by Pharmacist
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201511065RIND
Record Dates: First submitted 2016-02-11; First posted 2016-05-11 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Infection
Keywords: broad-spectrum antimicrobial; antibiotics pharmacist
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- inpatient under broad-spectrum antibiotics: medical review
  Interventions: Drug: medical review of controlled broad-spectrum antibiotics

INTERVENTIONS:
Drug: medical review of controlled broad-spectrum antibiotics — medical review of outcome of antibiotics stewardship by pharmacists and infectious disease physicians

SUMMARY:
To study the outcome of antibiotics stewardship

DETAILED DESCRIPTION:
Retrospective cohort study by medical review and evaluation of broad-spectrum antibiotics to determine how appropriately it was bing used.

ELIGIBILITY:
inclusion criteria:

* Inpatient with infectious disease and under broad-spectrum antibiotics

exclusion criteria:

* Poor prognosis was diagnosed or received conservative therapy only.

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the investigators randomly do medical chart review of patients received broad-spectrum antibiotics from their hospital systems.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
The percentage of appropriateness of empirical antibiotics choosing. | up to 8 weeks
  For example,the inappropriate of piperacillin-tazobactam as empirical therapy was numbers of participants with no risk factors of deep tissue infection or DM foot /Number of participants treated with piperacillin-tazobactam for soft tissue infection.
The percentage of appropriateness of de-escalation of therapy. | up to 8 weeks
  For example,continued piperacillin-tazobactam was seen to be inappropriate when microbiologic results and clinical status permit de-escalation.

SECONDARY OUTCOMES:
Number of adverse events of antibiotics were recorded. | up to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Chen Yang, master, Principal Investigator — National Taiwan University Hospital, Yun-Lin Branch
Locations (1):
- National Taiwan University Hospital, Douliu, Dou-Liou, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided